CLINICAL TRIAL: NCT01379885
Title: Childhood Immunization: Reducing Immunization Distress (RID) Using Multi-Modal Distraction
Brief Title: Reducing Immunization Distress (RID)
Acronym: RID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Estimated sample size not achieved due to decline in number of eligible patients and difficulty recruiting and retaining research staff.
Sponsor: University of California, San Francisco (Other)
Collaborators: Pediatric Medical Group (Unknown)
Responsible Party: Principal Investigator, Linda Franck, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCaliforniaSF
Record Dates: First submitted 2011-06-13; First posted 2011-06-23 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Pain
Keywords: Pain; immunization; distraction; hypnosis; injections; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard technique (Active Comparator): Children in the ST group will receive vapocoolant spray and arm gripping adjacent to the injection site performed by MA 1(immunizer). A second MA (MA 2) will perform the visual distraction by descending contralateral arm vibration using the massage instrument (buzzer).
  Interventions: Behavioral: Standard technique
- Parent participation technique (Experimental): The children in the PPT group will receive the same sequence, except that the parent/caregiver will administer the visual distraction rather than by MA2
  Interventions: Behavioral: Parent participation technique

INTERVENTIONS:
Behavioral: Standard technique — Children in the ST group will receive vapocoolant spray and arm gripping adjacent to the injection site performed by MA 1(immunizer). A second MA (MA 2) will perform the visual distraction by descending contralateral arm vibration using the massage instrument (buzzer).
  Arms: Standard technique
Behavioral: Parent participation technique — The children in the PPT group will receive the same sequence, except that the parent/caregiver will administer the visual distraction rather than by MA2
  Arms: Parent participation technique

SUMMARY:
The purpose of this study is to compare the effectiveness of a more feasible method for reducing the pain and distress of childhood immunization with the standard method in use at the Pediatric Medical Group. A secondary aim is to evaluate the impact of parental involvement on the parent and child satisfaction with the immunization experience.

Study Hypotheses: In the standard, pre-kindergarten, two- or three vaccine sequence, there will be no statistically significant group differences between PPT and ST with respect to:

1. Child self-reported pain using the Faces Pain Scale-Revised (FPS-R) scale13 (primary outcome);
2. Parent report of child pain using the FPS-R;
3. Observer-rated child distress and pain using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale14;
4. Parent and child satisfaction with pain management during immunization measured by a 5-point Likert type scales;
5. Time required for completion of immunization from initiation of ST or PPT to 2 minutes after completion of the last injection.

DETAILED DESCRIPTION:
Berberich and Landman conducted a randomized clinical trial demonstrating efficacy of a multimodal distraction technique to reduce immunization distress (RID) in 4-6 year old children receiving pre-kindergarten immunizations. Widespread implementation would require fewer steps and a reduction of personnel and the current study addresses the practical time and personnel limitations of the method. The current RID trial proposes a randomized design to compare our current method, the standard technique, (ST), with its minimally altered approach where arm gripping and rubbing adjacent to the injection site are to be performed by the medical assistant conducting the injection, substituting for the non-commercially available 'arm gripper'. Pressure and rubbing stimuli at injection sites are documented to be equally effective. The ST will be compared against the parental participation technique, (PPT), whereby the parent participates in the delivery of pain-relieving interventions in lieu of the second medical assistant. The primary aim of the present proposal is to compare the effectiveness of the more feasible PPT to the ST in reducing the pain and distress of childhood immunization. A secondary aim is to evaluate the impact of parental involvement on the parent and child satisfaction with the immunization experience.

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 4-6 years, scheduled to receive the standard pre-kindergarten immunizations. This consists of two injections: the Dtap (diphtheria, tetanus, acellular pertussis) and IPV (injectable polio vaccine) or three injections: DTAP, IPV and MMR (measles, mumps, rubella);
* With or without prior exposure to ST at PMG;
* English speaking subject and parents

Exclusion Criteria:

* Acute concurrent illness;
* Invasive procedures such as cannulation, venipuncture or urinary VCG in the preceding 6 months;
* Hospitalization or ED visit, within the prior 6 months;
* Chronic medical conditions requiring repeated painful interventions;
* Inability to respond age appropriately with verbal and written answers to questions, to pain scale measures, or to questionnaires;
* Refusal to be videotaped.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Child pain intensity | 2 minutes after completion of the immunization series.
  Child self-reported pain using the Faces Pain Scale-Revised (FPS-R) scale (primary outcome); Parent report of child pain using the FPS-R.

SECONDARY OUTCOMES:
Time for completion of immunization | From the start of the procedure to 2 minutes after completion of the immunization series.
  Time required for completion of immunization from initiation of ST or PPT to 2 minutes after completion of the last injection.
Child and parent satisfaction with procedure | 2 minutes after completion of the immunization series.
  Child and parent self-reported satisfaction with the procedure using a 5-item questionnaire developed specifically for the study.
Child pain intensity | Immediately before, and after injection in each arm.
  Observer-rated child distress and pain using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda Franck, RN,PhD, Principal Investigator — University of California, San Francisco; Ralph Berberich, MD, Principal Investigator — Pediatric Medical Group
Locations (1):
- Pediatric Medical Group, Berkeley, California, United States

REFERENCES:
- [Background] Reis EC, Roth EK, Syphan JL, Tarbell SE, Holubkov R. Effective pain reduction for multiple immunization injections in young infants. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1115-20. doi: 10.1001/archpedi.157.11.1115. PMID 14609903
- [Background] Taddio A, Chambers CT, Halperin SA, Ipp M, Lockett D, Rieder MJ, Shah V. Inadequate pain management during routine childhood immunizations: the nerve of it. Clin Ther. 2009;31 Suppl 2:S152-67. doi: 10.1016/j.clinthera.2009.07.022. PMID 19781434
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline (summary). CMAJ. 2010 Dec 14;182(18):1989-95. doi: 10.1503/cmaj.092048. Epub 2010 Nov 22. No abstract available. PMID 21098067
- [Background] Hamilton JG. Needle phobia: a neglected diagnosis. J Fam Pract. 1995 Aug;41(2):169-75. PMID 7636457
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline. CMAJ. 2010 Dec 14;182(18):E843-55. doi: 10.1503/cmaj.101720. Epub 2010 Nov 22. No abstract available. PMID 21098062
- [Background] Taddio A, Manley J, Potash L, Ipp M, Sgro M, Shah V. Routine immunization practices: use of topical anesthetics and oral analgesics. Pediatrics. 2007 Sep;120(3):e637-43. doi: 10.1542/peds.2006-3351. PMID 17766503
- [Background] Parvez E, Stinson J, Boon H, Goldman J, Shah V, Taddio A. Mothers' beliefs about analgesia during childhood immunization. Paediatr Child Health. 2010 May;15(5):289-93. doi: 10.1093/pch/15.5.289. PMID 21532793
- [Background] Schechter NL, Bernstein BA, Zempsky WT, Bright NS, Willard AK. Educational outreach to reduce immunization pain in office settings. Pediatrics. 2010 Dec;126(6):e1514-21. doi: 10.1542/peds.2010-1597. Epub 2010 Nov 15. PMID 21078736
- [Background] Berberich FR, Landman Z. Reducing immunization discomfort in 4- to 6-year-old children: a randomized clinical trial. Pediatrics. 2009 Aug;124(2):e203-9. doi: 10.1542/peds.2007-3466. Epub 2009 Jul 13. PMID 19596729
- [Background] Barnhill BJ, Holbert MD, Jackson NM, Erickson RS. Using pressure to decrease the pain of intramuscular injections. J Pain Symptom Manage. 1996 Jul;12(1):52-8. doi: 10.1016/0885-3924(96)00049-8. PMID 8718917
- [Background] Chung JW, Ng WM, Wong TK. An experimental study on the use of manual pressure to reduce pain in intramuscular injections. J Clin Nurs. 2002 Jul;11(4):457-61. doi: 10.1046/j.1365-2702.2002.00645.x. PMID 12100641
- [Background] Taddio A, Lord A, Hogan ME, Kikuta A, Yiu A, Darra E, Bruinse B, Keogh T, Stephens D. A randomized controlled trial of analgesia during vaccination in adults. Vaccine. 2010 Jul 19;28(32):5365-9. doi: 10.1016/j.vaccine.2010.05.015. Epub 2010 May 16. PMID 20483194
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Derived] Franck LS, Berberich FR, Taddio A. Parent participation in a childhood immunization pain reduction method. Clin Pediatr (Phila). 2015 Mar;54(3):228-35. doi: 10.1177/0009922814561593. Epub 2014 Dec 3. PMID 25475591